CLINICAL TRIAL: NCT05715918
Title: Double-blind, Placebo-controlled, Randomized Study of Tolerability, Safety and Immunogenicity of the Inactivated Whole-virion Concentrated Purified Coronavirus Vaccine, Produced by FSBSI "Chumakov Federal Scientific Center for Research and Development of Immune-and-Biological Products", of Children at the Age of 12-17 Years Inclusive"
Brief Title: Double-blind, Placebo-controlled, Randomized Study of the Tolerability, Safety and Immunogenicity of an Inactivated Whole Virion Concentrated Purified Vaccine (CoviVac) Against Covid-19 of Children at the Age of 12-17 Years Inclusive"
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chumakov Federal Scientific Center for Research and Development of Immune-and-Biological Products (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: № VKI-D-III-12/21
Record Dates: First submitted 2023-02-06; First posted 2023-02-08 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Vaccine
Keywords: COVID-19; Coronavirus infections; Vaccine; SARS-CoV-2; Immunobiological medicine
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Vaccines; Injections, Intramuscular

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine (Experimental): Group 1 - 150 volunteers, Vaccine 0.5 ml, 21 days interval, post-vaccination observation period of 21 days.
  An additional objective of the study is to evaluate the safety, immunogenicity and efficacy of the CoviVac vaccine in the period from 21 days to 24 weeks after the second vaccination in comparison with placebo throughout the study.
  Interventions: Biological: Vaccine for intramuscular injection
- Placebo (Placebo Comparator): No active ingredient in the placebo
  Group 2 - 150 volunteers, Placebo 0.5 ml, 21 days interval, post-vaccination observation period of 21 days.
  An additional objective of the study is to evaluate the safety, immunogenicity and efficacy of the CoviVac vaccine in the period from 21 days to 24 weeks after the second vaccination in comparison with placebo throughout the study.
  Interventions: Other: Placebo comparator (without active ingredient) for intramuscular injection

INTERVENTIONS:
Biological: Vaccine for intramuscular injection — Volunteers ( Group 1 - 150) will receive the vaccine twice spaced 21 days apart, intramuscularly, at a dose of 0.5 ml
  Arms: Vaccine
Other: Placebo comparator (without active ingredient) for intramuscular injection — Volunteers ( Group 2 - 150) will receive the vaccine twice spaced 21 days apart, intramuscularly, at a dose of 0.5 ml
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo controlled, multi-center clinical trials of the tolerability, safety and immunogenicity of the inactivated whole-virion concentrated purified vaccine against COVID-19, manufactured by FSBSI "Chumakov FSC R&D IBP RAS", of childrens aged 12-17" (Clinical trials, phase III). Study purpose is to assess the tolerability, safety and immunogenicity of the inactivated whole-virion concentrated purified coronavirus vaccine of chidrens aged 12-17

DETAILED DESCRIPTION:
Recruitment of volunteers will be competitive. A maximum of 450 children aged 12 to 17 years inclusive will be screened in the study, of which it is planned to include and randomize 300 children who meet the criteria for inclusion in the study and do not have non-inclusion criteria, data on which will be used for subsequent safety and immunogenicity analysis.

Group 1 - 150 volunteers who will be vaccinated with the Nobivac vaccine twice with an interval of 21 days intramuscularly.

Group 2 - 150 volunteers who will receive a placebo twice with an interval of 21 days intramuscularly.

In case of withdrawal of volunteers from the study, their replacement is not provided.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must meet the following inclusion criteria:

Type of participants • Healthy volunteers.

Age at the time of signing the Informed Consent

• from 12 to 17 years inclusive (12 years 0 months 0 days - 17 years 11 months 30 days).

Paul • Male or female.

Reproductive characteristics

* For girls with a history of mensis - a negative pregnancy test and consent to adhere to adequate methods of contraception (use of contraceptives within a month after the second vaccination). Girls should use methods of contraception with a reliability of more than 90% (cervical caps with spermicide, diaphragms with spermicide, condoms, intrauterine spirals).
* For young men capable of conception - consent to adhere to adequate methods of contraception (use of contraceptives within a month after the second vaccination). Young men and their sexual partners should use methods of contraception with a reliability of more than 90% (cervical caps with spermicide, diaphragms with spermicide, condoms, intrauterine spirals).

Research procedures

* Written Informed consent of a volunteer (14 years and older) and one of the parents to participate in a clinical trial.
* Volunteers who are able to fulfill Protocol requirements (i.e. answer phone calls, fill out a Self-observation Diary, come to control visits).

Non-inclusion criteria:

* Volunteers cannot be included in the study if any of the following criteria are present:

SARS-CoV-2 infection

* A case of established COVID-19 disease confirmed by PCR and/or ELISA in the last 6 months.
* History of contacts with confirmed or suspected cases of SARS-CoV-2 infection within 14 days prior to vaccination.
* Positive IgM or IgG to SARS-CoV-2 detected on Screening.
* Positive PCR test for SARS-CoV-2 at Screening / before vaccination.

Diseases or medical conditions

* Serious post-vaccination reaction (temperature above 40 C, hyperemia or edema more than 8 cm in diameter) or complication (collapse or shock-like condition that developed within 48 hours after vaccination; convulsions, accompanied or not accompanied by a feverish state) to any previous vaccination.
* Burdened allergic history (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, serum sickness in the anamnesis, hypersensitivity or allergic reactions to the introduction of any vaccines in the anamnesis, known allergic reactions to vaccine components, etc.).
* Guillain-Barre syndrome (acute polyradiculitis) in the anamnesis.
* The axillary temperature at the time of vaccination is more than 37.0 ° C.
* Positive blood test for HIV, syphilis, hepatitis B/C.
* Acute infectious diseases (recovery earl

Exclusion Criteria:

- • Withdrawal of Informed consent by a volunteer and/or a parent of a volunteer;

* The volunteer was included in violation of the inclusion/non-inclusion criteria of the Protocol;
* Availability of inclusion/non-inclusion criteria before vaccination;
* Any condition of a volunteer that requires, in the reasoned opinion of a medical researcher, the withdrawal of a volunteer from the study;
* The established fact of pregnancy before the second vaccination;
* Taking unauthorized medications (see section 6.2);
* The volunteer's incompetence with the study procedures;
* The volunteer refuses to cooperate or is undisciplined (for example, failure to attend a scheduled visit without warning the researcher and/or loss of communication with the volunteer), or dropped out of observation;
* For administrative reasons (termination of the study by the Sponsor or regulatory authorities), as well as in case of gross violations of the protocol that may affect the results of the study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) | 21 days
  The percentage of volunteers with an increase in geometric mean titer of specific antibodies (GMT) on day 21 after the second dose of vaccine / placebo in the virus neutralization test and ELISA.
Geometric mean titer (GMT) | 21 days
  The multiplicity of the increase in the geometric mean titer of specific antibodies (GMT) for 21 days after the second vaccination in the viral neutralization reaction and ELISA reaction.
The level of seroconversion | 21 days
  The level of seroconversion (titer of specific antibodies ≥ 4 times) on 21 days after the second vaccination in the reaction of virusneutralization and ELISA reaction

SECONDARY OUTCOMES:
Geometric mean titer (GMT) | 24 weeks
  The mean geometric titer of specific antibodies (GMT) 12 and 24 weeks after the second vaccination in the viral neutralization reaction and ELISA reaction.
Geometric mean titer (GMT) | 24 weeks
  The multiplicity of the increase in the geometric mean titer of specific antibodies (GMT) 12 and 24 weeks after the second vaccination in the viral neutralization reaction and ELISA reaction.
The level of seroconversion | 24 weeks
  The level of seroconversion (titer of specific antibodies ≥ 4 times) 12 and 24 weeks after the second vaccination in the viral neutralization reaction and ELISA reaction.

CONTACTS AND LOCATIONS:
Locations (4):
- Russia (4):
  - State Budgetary Health Institution of the Moscow Region "Elektrostal Central City Hospital", Elektrostal, Moscow
  - Kirov Regional State Budgetary Health Institution "Kirov Regional Children's Clinical Hospital", Kirov
  - FSBSI Chumakov FSC R&D IBP RAS, Moscow
  - St. Petersburg State Budgetary Health Institution "Children's City Polyclinic No. 45 of the Nevsky District", Saint Petersburg